CLINICAL TRIAL: NCT06952673
Title: Study on the 'Seismocardiography-Electrocardiography' Coupling Dynamics and Its Exercise-load Reactivity Model in Healthy Individuals
Brief Title: Study on Multi-Modality Models of Cardiac Function in Healthy Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ruiwei Digital Technology Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RW-H-001
Record Dates: First submitted 2025-04-19; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers Only
Keywords: Seismocardiography, ECG, Exercise Responsivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multiple speed increments on a treadmill for healthy individuals (Experimental): Healthy participants will undergo the following experimental protocol: After wearing microsensors and a respiratory/metabolic testing mask, they will rest quietly for 3 minutes, then begin walking at a speed of 3 km/h for 6 minutes, followed by a 3-minute quiet rest period. This will be followed by walking at 4 km/h for 6 minutes and another 3-minute rest. The protocol continues with subsequent stages at progressively increasing speeds of 5 km/h, 6 km/h, 7 km/h, and 8 km/h, each involving 6 minutes of walking followed by 3 minutes of rest.
  Interventions: Behavioral: Multiple speed increments from 3km/h to 8km/h on a treadmill

INTERVENTIONS:
Behavioral: Multiple speed increments from 3km/h to 8km/h on a treadmill — Healthy participants will undergo a fixed experimental protocol of multi-stage treadmill speed walking/running wearing microsensors and a respiratory/metabolic testing mask.

SUMMARY:
In this study, wearable multi-modal microsensors were deployed to simultaneously capture seismocardiography (SCG) and electrocardiography (ECG) signals, delineating the exercise-load-dependent responsiveness of SCG-ECG dynamic coupling during graded-speed treadmill protocols.

DETAILED DESCRIPTION:
The heart adapts to varying exercise loads primarily by augmenting heart rate and contractility to achieve matching increases in cardiac output. However, whether there exists an intrinsic triaxial regulatory mechanism governing the interdependencies among 'exercise load - heart rate response - contractility response' remains unknown. In this study, participants performed treadmill exercise at multiple speed gradients (3-8 km/h). Seismocardiography (SCG) signals were captured via an inertial measurement unit (IMU) positioned on the precordium and were used to characterize mechanical cardiac contractility. Single-lead precordial ECG provided heart rate dynamics, while CPET-derived oxygen uptake (VO₂) indexed exercise intensity. The primary objectives were to delineate SCG-ECG responsivity patterns under graded exercise intensities and quantify potential intrinsic laws linking exercise load, heart rate adaptation, and contractility modulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Healthy individuals with no significant medical history
* Signed informed consent as an acceptance to participate to the trial

Exclusion Criteria:

* History of severe cardiovascular, cerebrovascular, pulmonary, hepatic, renal, psychiatric, or other critical systemic disorders
* Peripheral vascular diseases, musculoskeletal disorders, or other conditions limiting physical mobility
* Uncontrolled hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg)
* History of anemia
* Moderate to severe obesity (BMI ≥32.5 kg/m²)
* Pregnant or lactating women
* Any other conditions deemed ineligible for participation per investigator's discretion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in SCG features (amplitude in m/s²) | The entire test will be completed in approximately 90 minutes.
  Triaxial accelerometer-derived SCG signals (500 Hz) yielded peak-to-peak amplitudes (m/s²) per cardiac cycle and values were averaged over rest artifact-free 30-second epochs.

SECONDARY OUTCOMES:
Changes in ECG features (R-R interval in ms) | The entire test will be completed in approximately 90 minutes.
  R-R intervals (ms) were computed from single lead ECG (250 Hz) and auto-detected R-peaks were confirmed by amplitude and slope thresholds. R-R intervals were averaged over hardware synchronized SCG 30-second epochs.